CLINICAL TRIAL: NCT00306527
Title: A Phase III, Observer-Blind, Randomized, Multi-Center Study to Evaluate Safety, Tolerability and Immunogenicity (in a Subset) Following a Single Intramuscular Dose of a Trivalent Subunit Influenza Vaccine Produced Either in Mammalian Cell Culture or in Embryonated Hen Eggs, in Healthy Adult and Elderly Subjects Who Received Either One or the Other Vaccine One Year Before in the V58P4 Study.
Brief Title: Comparison of Safety, Tolerability and Immunogenicity of Influenza Vaccines in Adults and Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis Vaccines and Diagnostics S.r.l. (Unknown)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: V58P4E1; EUDRACT: 2005-001902-26
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Results first posted 2013-01-11 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Influenza
Keywords: Influenza; adult/elderly; flu cell culture; vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (8):
- cTIV\cTIV (adults) (Active Comparator): Subjects (18-60 years of age) previously vaccinated with cell-derived influenza vaccine (cTIV), received one dose of cell-derived trivalent influenza vaccine (cTIV) one year later, in this study.
  Interventions: Biological: Cell culture derived influenza vaccine
- cTIV\TIV (adults) (Active Comparator): Subjects (18-60 years of age) previously vaccinated with cell-derived influenza vaccine (cTIV), received one dose of an egg-derived trivalent influenza vaccine (TIV) one year later, in this study.
  Interventions: Biological: egg-derived influenza subunit vaccine
- cTIV\cTIV (elderly) (Active Comparator): Subjects (≥61 years of age) previously vaccinated with cell-derived influenza vaccine (cTIV), received one dose of cell-derived trivalent influenza vaccine (cTIV) one year later, in this study.
  Interventions: Biological: Cell culture derived influenza vaccine
- cTIV\TIV (elderly) (Active Comparator): Subjects (≥61years of age) previously vaccinated with cell-derived influenza vaccine (cTIV), received one dose of an egg-derived trivalent influenza vaccine (TIV) one year later, in this study.
  Interventions: Biological: egg-derived influenza subunit vaccine
- TIV\TIV (adults) (Active Comparator): Subjects (18-60 years of age) previously vaccinated with egg-derived influenza vaccine (TIV), received one dose of egg-derived trivalent influenza vaccine (TIV) one year later, in this study.
  Interventions: Biological: egg-derived influenza subunit vaccine
- TIV\cTIV (adults) (Active Comparator): Subjects (18-60 years of age) previously vaccinated with egg-derived influenza vaccine (TIV), received one dose of cell-derived trivalent influenza (cTIV) one year later, in this study.
  Interventions: Biological: Cell culture derived influenza vaccine
- TIV\TIV (elderly) (Active Comparator): Subjects (≥61 years of age) previously vaccinated with egg-derived influenza vaccine (TIV), received one dose of egg-derived trivalent influenza vaccine (TIV) one year later, in this study.
  Interventions: Biological: egg-derived influenza subunit vaccine
- TIV\cTIV (elderly) (Active Comparator): Subjects (≥61 years of age) previously vaccinated with egg-derived influenza vaccine (TIV), received one dose of cell-derived trivalent influenza (cTIV) one year later, in this study.
  Interventions: Biological: Cell culture derived influenza vaccine

INTERVENTIONS:
Biological: Cell culture derived influenza vaccine — as a single IM injection of 0.5 ml in the deltoid muscle, preferably of the non-dominant arm
  Arms: TIV\cTIV (adults); TIV\cTIV (elderly); cTIV\cTIV (adults); cTIV\cTIV (elderly)
Biological: egg-derived influenza subunit vaccine — as a single IM injection of 0.5 ml in the deltoid muscle, preferably of the non-dominant arm
  Arms: TIV\TIV (adults); TIV\TIV (elderly); cTIV\TIV (adults); cTIV\TIV (elderly)

SUMMARY:
The purpose of the study is to evaluate safety, tolerability and immunogenicity (in a subset) following a dose of a trivalent subunit influenza vaccine produced either in mammalian cells or in embryonated hen eggs, in healthy adult and elderly subjects who received either vaccine one year before (2004) in the study V58P4.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to < 61 years of age (first age group) OR 61 years of age and older (second age group) at enrolment in V58P4
2. Mentally competent to understand the nature, the scope and the consequences of the study
3. Able and willing to give written informed consent prior to study entry
4. Available for all the visits scheduled in the study
5. in good health as determined by:

   1. Medical history related to the previous six months,
   2. Physical examination,
   3. Clinical judgment of the investigator.

Exclusion Criteria:

1. Unwilling or unable to give written informed consent to participate in the study
2. Currently experiencing an acute infectious disease
3. Any serious disease such as, for example:

   1. Cancer (except for benign or localized skin cancer and non metastatic prostate cancer not currently treated with chemotherapy)
   2. Autoimmune disease (including rheumatoid arthritis)
   3. Advanced arteriosclerotic disease or complicated diabetes mellitus
   4. Chronic obstructive pulmonary disease (COPD) requiring oxygen therapy
   5. Acute or progressive hepatic disease
   6. Acute or progressive renal disease
   7. Congestive heart failure
4. Surgery planned during the study period
5. Bleeding diathesis
6. History of hypersensitivity to any component of the study medication or chemically related substances, such as allergy to eggs or egg products
7. Known or suspected impairment/alteration of immune function resulting from:

   1. Receipt of immunosuppressive therapy (any cortical steroid or cancer chemotherapy)
   2. Receipt of immunostimulants
   3. Receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the past 3 months and for the full length of the study
   4. High risk for developing an immunocompromising disease
8. History of drug or alcohol abuse
9. Laboratory confirmed influenza disease in the past 6 months
10. Received influenza vaccine within the past 6 months
11. Received another vaccine or any investigational agent within the past 60 days, or expect to receive another vaccine within 3 weeks following the study vaccination
12. Participation in another clinical trial within 90 days prior to enrollment and throughout the full length of the study
13. Any acute respiratory disease or infections requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis is acceptable) or experienced fever _ 38°C within the past 5 days
14. Pregnant/ breast feeding women or women who refuse to use a reliable contraceptive method during the first three weeks after vaccination
15. Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2235 (Actual)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (5):
- Poland (5):
  - Wojewódzki Szpital Dzieci_cy, Ul. Langiewicza 2, Kielce
  - Centrum Bada_ Farmakologii Klinicznej, Ul. Ujastek 3, Krakow
  - NZOZ Jagiello_skie, Centrum Medyczne Sp. Z O.o., O_. Jagiello_skie 1, Kraków
  - NZOZ Praktyka Grupowa Lekarzy Rodzinnych, "Familia" Sp. z o.o., Pl. Sikorskiego 6a, Kraków
  - Szpital Jana Pawła II, Oddz. Neuroinfekcji, Ul. Pr_dnicka 80, Kraków

REFERENCES:
- [Result] Szymczakiewicz-Multanowska A, Lattanzi M, Izu A, Casula D, Sparacio M, Kovacs C, Groth N. Safety assessment and immunogenicity of a cell-culture-derived influenza vaccine in adults and elderly subjects over three successive influenza seasons. Hum Vaccin Immunother. 2012 May;8(5):645-52. doi: 10.4161/hv.19493. Epub 2012 May 1. PMID 22418809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 5 study centers in Poland.
Pre-assignment Details: All subjects enrolled were included in the trial.
Groups:
- Adults (cTIV\cTIV) + (TIV\cTIV): Subjects (18-60 years of age) who previously received one dose of either cell-derived (cTIV) or egg derived (TIV) trivalent influenza vaccine received one dose of cTIV in this study, one year later.
- Adults (cTIV\TIV) + (TIV\TIV): Subjects (18-60 years of age) who previously received one dose of either cell-derived (cTIV) or egg derived (TIV) trivalent influenza vaccine received one dose of TIV in this study, one year later.
- Elderly (cTIV\cTIV) + (TIV\cTIV): Subjects(≥61years of age ) who previously received one dose of either cell-derived (cTIV) or egg derived (TIV) trivalent influenza vaccine received one dose of cTIV in this study, one year later.
- Elderly (cTIV\TIV) + (TIV\TIV): Subjects (≥61years) who previously received one dose of either cell-derived (cTIV) or egg derived (TIV) trivalent influenza vaccine received one dose of TIV in this study, one year later.
Period: Overall Study
Arm/Group | Adults (cTIV\cTIV) + (TIV\cTIV) | Adults (cTIV\TIV) + (TIV\TIV) | Elderly (cTIV\cTIV) + (TIV\cTIV) | Elderly (cTIV\TIV) + (TIV\TIV)
Started | 533 | 534 | 572 | 596
Completed | 527 | 527 | 567 (3 of 4 deaths in the elderly subjects resulted in premature discontinuation. Refer to OM2 .) | 590
Not Completed | 6 | 7 | 5 | 6
Not completed — Lost to Follow-up | 3 | 4 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Death | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Adults (cTIV\cTIV) + (TIV\cTIV): Subjects(18-60 years of age) who previously received one dose of either cell-derived (cTIV) or egg derived (TIV) trivalent influenza vaccine, received one dose of cTIV in this study, one year later.
- Elderly (cTIV\cTIV) + (TIV\cTIV): Subjects(≥61 years of age) who previously received one dose of either cell-derived (cTIV) or egg derived (TIV) trivalent influenza vaccine, received one dose of cTIV in this study, one year later.
- Elderly (cTIV\TIV) + (TIV\TIV): Subjects (≥61 years of age) who previously received one dose of either cell-derived (cTIV) or egg derived (TIV) trivalent influenza vaccine received one dose of TIV in this study, one year later.
- Total: Total of all reporting groups
Arm/Group | Adults (cTIV\cTIV) + (TIV\cTIV) | Elderly (cTIV\cTIV) + (TIV\cTIV) | Adults (cTIV\TIV) + (TIV\TIV) | Elderly (cTIV\TIV) + (TIV\TIV) | Total
Number analyzed (Participants) | 533 | 572 | 534 | 596 | 2235
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (12.7) | 69.2 (5.7) | 39.0 (12.5) | 69.9 (5.7) | 55.2 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 308 | 309 | 353 | 1278
  Male | 225 | 264 | 225 | 243 | 957

OUTCOME MEASURES:

1. Secondary Outcome: Six-months Safety Data of Subjects After One Dose of Cell Culture Derived or Egg-derived Influenza Vaccine
Description: To collect additional safety data for 6 months after vaccination with one dose of cell culture derived or egg-derived influenza vaccine in terms of serious adverse events (SAEs), adverse events (AEs) necessitating a physician's visit and/or resulting in premature subject's withdrawal from study.
Time Frame: Up to 6 months postvaccination
Population: This analysis was done on the safety dataset.
Measure: Number; unit: Participants
Groups:
- cTIV\cTIV (Elderly): Subjects (≥61years of age) previously vaccinated with cell-derived influenza vaccine (cTIV), received one dose of cell-derived trivalent influenza vaccine (cTIV) one year later, in this study.
- TIV\TIV (Elderly): Subjects (≥61years of age) previously vaccinated with egg-derived influenza vaccine (TIV), received one dose of egg-derived trivalent influenza vaccine (TIV) one year later, in this study.
- TIV\cTIV (Elderly): Subjects (≥61years of age) previously vaccinated with egg-derived influenza vaccine (TIV), received one dose of cell-derived trivalent influenza (cTIV) one year later, in this study.
Arm/Group | cTIV\cTIV (Adults) | cTIV\TIV (Adults) | cTIV\cTIV (Elderly) | cTIV\TIV (Elderly) | TIV\TIV (Adults) | TIV\cTIV (Adults) | TIV\TIV (Elderly) | TIV\cTIV (Elderly)
Number analyzed (Participants) | 272 | 274 | 290 | 297 | 260 | 261 | 300 | 281
Participants
  Any AE | 50 | 38 | 70 | 58 | 35 | 44 | 67 | 76
  At least possibly related AE | 2 | 4 | 2 | 5 | 2 | 4 | 2 | 5
  Any SAE | 5 | 4 | 13 | 13 | 0 | 4 | 17 | 10
  At least possibly related SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any death | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2

2. Secondary Outcome: Geometric Mean Titers (GMTs) After One Dose of Cell Culture-derived or the Egg-derived Influenza Vaccine in Adult and Elderly Subjects
Description: The haemagglutinin inhibition (HI) antibody titer response following one 0.5 mL dose of either cell derived (cTIV) or egg-derived vaccine (TIV) in adult and elderly subjects is reported as GMTs.
  The HI GMTs were evaluated using egg-derived antigen assay.
Time Frame: Day 22 postvaccination
Population: The analysis was done on the immunogenicity subset.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | cTIV\cTIV (Adults) | cTIV\TIV (Adults) | cTIV\cTIV (Elderly) | cTIV\TIV (Elderly) | TIV\TIV (Adults) | TIV\cTIV (Adults) | TIV\TIV (Elderly) | TIV\cTIV (Elderly)
Number analyzed (Participants) | 60 | 60 | 61 | 61 | 59 | 60 | 61 | 61
Titers
  A/H1N1 strain (Day 1) | 40 [28 to 58] | 34 [24 to 48] | 26 [19 to 35] | 20 [15 to 27] | 35 [25 to 51] | 36 [25 to 51] | 24 [18 to 32] | 26 [19 to 35]
  A/H1N1 strain (Day 22) | 87 [65 to 116] | 83 [62 to 111] | 57 [43 to 76] | 61 [46 to 80] | 72 [53 to 96] | 104 [78 to 140] | 61 [46 to 81] | 80 [61 to 106]
  A/H3N2 strain (Day 1) | 16 [12 to 21] | 18 [13 to 23] | 20 [15 to 26] | 26 [19 to 34] | 19 [15 to 25] | 21 [16 to 28] | 19 [14 to 25] | 20 [15 to 27]
  A/H3N2 strain (Day 22) | 173 [129 to 233] | 109 [81 to 146] | 229 [163 to 321] | 197 [141 to 277] | 78 [58 to 105] | 170 [127 to 229] | 125 [89 to 175] | 251 [178 to 352]
  B strain (Day 1) | 30 [22 to 40] | 26 [19 to 35] | 36 [27 to 48] | 48 [36 to 64] | 37 [27 to 50] | 35 [26 to 48] | 26 [19 to 34] | 37 [27 to 49]
  B strain (Day 22) | 77 [60 to 99] | 71 [55 to 91] | 84 [64 to 111] | 128 [97 to 168] | 67 [52 to 86] | 104 [81 to 133] | 68 [51 to 89] | 116 [88 to 154]

3. Secondary Outcome: Geometric Mean Ratios (GMRs), After One Dose of the Cell Culture-derived or the Egg-derived Influenza Vaccine in Adult and Elderly Subjects
Description: Immunogenicity was assessed in terms of GMR in adult and elderly subjects following one 0.5ml dose of either the cTIV vaccine or the TIV vaccine, according to the CHMP criteria.
  The European licensure (CHMP) criteria was met if the mean geometric increase (GMR, day 22/day 1) in HI antibody titer is >2.5 for adults and >2.0 for elderly subjects.
Time Frame: Day 22 postvaccination
Population: The analysis was done on the immunogenicity subset.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | cTIV\cTIV (Adults) | cTIV\TIV (Adults) | cTIV\cTIV (Elderly) | cTIV\TIV (Elderly) | TIV\TIV (Adults) | TIV\cTIV (Adults) | TIV\TIV (Elderly) | TIV\cTIV (Elderly)
Number analyzed (Participants) | 60 | 60 | 61 | 61 | 59 | 60 | 61 | 61
Ratio
  A/H1N1 strain | 2.14 [1.67 to 2.74] | 2.46 [1.92 to 3.15] | 2.2 [1.71 to 2.84] | 2.98 [2.31 to 3.84] | 2.02 [1.58 to 2.6] | 2.91 [2.27 to 3.73] | 2.54 [1.97 to 3.28] | 3.11 [2.41 to 4.02]
  A/H3N2 strain | 11 [8.13 to 14] | 6.17 [4.64 to 8.2] | 12 [8.49 to 16] | 7.64 [5.58 to 10] | 4.09 [3.07 to 5.45] | 8.05 [6.06 to 11] | 6.59 [4.81 to 9.04] | 12 [8.94 to 17]
  B strain | 2.61 [2.07 to 3.29] | 2.7 [2.14 to 3.41] | 2.37 [1.86 to 3.03] | 2.67 [2.09 to 3.42] | 1.81 [1.43 to 2.29] | 2.93 [2.32 to 3.7] | 2.64 [2.07 to 3.38] | 3.19 [2.5 to 4.07]

4. Secondary Outcome: Percentages of Adult and Elderly Subjects Achieving HI Titers ≥ 40 After One Dose of the Cell Culture-derived or the Egg-derived Influenza Vaccine.
Description: Immunogenicity was assessed in terms of percentages of adult and elderly subjects achieving HI titers≥40,after one dose of either the cTIV vaccine or the TIV vaccine.
  European (CHMP) criteria is met if the percentage of subjects achieving HI titers ≥ 40 is > 70% for adults and >60% for elderly.
Time Frame: Day 22 postvaccination
Population: This analysis was done on immunogenicity subset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | cTIV\cTIV (Adults) | cTIV\TIV (Adults) | cTIV\cTIV (Elderly) | cTIV\TIV (Elderly) | TIV\TIV (Adults) | TIV\cTIV (Adults) | TIV\TIV (Elderly) | TIV\cTIV (Elderly)
Number analyzed (Participants) | 60 | 60 | 61 | 61 | 59 | 60 | 61 | 61
Percentages of subjects
  A/H1N1 strain (Day 1) | 57 [43 to 69] | 48 [35 to 62] | 49 [36 to 62] | 36 [24 to 49] | 54 [41 to 67] | 57 [43 to 69] | 36 [24 to 49] | 48 [35 to 61]
  A/H1N1 strain (Day 22) | 85 [73 to 93] | 80 [68 to 89] | 77 [65 to 87] | 74 [61 to 84] | 80 [67 to 89] | 90 [79 to 96] | 69 [56 to 80] | 82 [70 to 91]
  A/H3N2 strain (Day 1) | 25 [15 to 38] | 27 [16 to 40] | 30 [19 to 43] | 39 [27 to 53] | 32 [21 to 46] | 33 [22 to 47] | 26 [16 to 39] | 34 [23 to 48]
  A/H3N2 strain (Day 22) | 92 [82 to 97] | 95 [86 to 99] | 97 [89 to 100] | 95 [86 to 99] | 86 [75 to 94] | 92 [82 to 97] | 87 [76 to 94] | 92 [82 to 97]
  B strain (Day 1) | 50 [37 to 63] | 50 [37 to 63] | 59 [46 to 71] | 61 [47 to 73] | 54 [41 to 67] | 58 [45 to 71] | 43 [30 to 56] | 62 [49 to 74]
  B strain (Day 22) | 80 [68 to 89] | 90 [79 to 96] | 84 [72 to 92] | 92 [82 to 97] | 85 [73 to 93] | 87 [75 to 94] | 84 [72 to 92] | 90 [80 to 96]

5. Secondary Outcome: Percentages of Adult and Elderly Subjects With Seroconversion or Significant Increase in HI Antibody Titers After One Dose of Cell Culture-derived or the Egg-derived Influenza Vaccine.
Description: Immunogenicity was assessed in terms of percentages of adult and elderly subjects showing seroconversion or significant increase in HI antibody titers after one dose of cell culture-derived or the egg-derived influenza vaccine.
  Seroconversion or significant increase as per European Licensure (CHMP) criteria is defined as percentage of subjects with a prevaccination HI titer <10 to a postvaccination titer ≥ 40 for adults and ≥ 30 for elderly. Significant increase is defined as percentage of subjects with a prevaccination HI titer ≥ 10 and a ≥ 4-fold increase in postvaccination HI antibody titer.
Time Frame: Day 22 postvaccination
Population: This analysis was done on the immunogenicity subset.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | cTIV\cTIV (Adults) | cTIV\TIV (Adults) | cTIV\cTIV (Elderly) | cTIV\TIV (Elderly) | TIV\TIV (Adults) | TIV\cTIV (Adults) | TIV\TIV (Elderly) | TIV\cTIV (Elderly)
Number analyzed (Participants) | 60 | 60 | 61 | 61 | 59 | 60 | 61 | 61
Percentages of subjects
  A/H1N1 strain | 22 [12 to 34] | 32 [20 to 45] | 30 [19 to 43] | 34 [23 to 48] | 24 [14 to 37] | 30 [19 to 43] | 30 [19 to 43] | 43 [30 to 56]
  A/H3N2 strain | 82 [70 to 90] | 85 [73 to 93] | 84 [72 to 92] | 80 [68 to 89] | 61 [47 to 73] | 80 [68 to 89] | 77 [65 to 87] | 82 [70 to 91]
  B strain | 28 [17 to 41] | 33 [22 to 47] | 28 [17 to 41] | 34 [23 to 48] | 27 [16 to 40] | 40 [28 to 53] | 31 [20 to 44] | 41 [29 to 54]

6. Primary Outcome: Number of Subjects Reporting Solicited Adverse Events After One Dose of Cell Culture-derived or the Egg-derived Influenza Vaccine
Description: To assess the safety and tolerability in terms of number of adult and elderly subjects reporting solicited adverse events following one dose of the cTIV or the TIV vaccine .
Time Frame: Day 1 to Day 7 postvaccination
Population: This analysis was done on safety dataset
Measure: Number; unit: Participants
Arm/Group | cTIV\cTIV (Adults) | cTIV\TIV (Adults) | cTIV\cTIV (Elderly) | cTIV\TIV (Elderly) | TIV\TIV (Adults) | TIV\cTIV (Adults) | TIV\TIV (Elderly) | TIV\cTIV (Elderly)
Number analyzed (Participants) | 272 | 274 | 290 | 297 | 260 | 261 | 300 | 281
Participants
  Local | 78 | 73 | 47 | 51 | 76 | 84 | 47 | 55
  Injection site ecchymosis | 13 | 11 | 12 | 15 | 13 | 13 | 18 | 11
  Injection site erythema | 32 | 26 | 22 | 19 | 40 | 27 | 16 | 24
  Injection site induration | 17 | 11 | 10 | 7 | 20 | 18 | 10 | 14
  Injection site swelling | 8 | 4 | 7 | 5 | 12 | 9 | 4 | 8
  Injection site pain | 52 | 45 | 22 | 21 | 46 | 63 | 19 | 26
  Systemic | 41 | 46 | 37 | 40 | 42 | 46 | 37 | 47
  Chills | 7 | 4 | 8 | 7 | 4 | 8 | 5 | 10
  Malaise | 20 | 18 | 19 | 19 | 20 | 27 | 20 | 29
  Myalgia | 19 | 20 | 13 | 9 | 22 | 19 | 10 | 21
  Arthralgia | 10 | 7 | 14 | 14 | 9 | 11 | 11 | 15
  Headache | 24 | 21 | 16 | 22 | 21 | 27 | 15 | 20
  Sweat | 10 | 8 | 10 | 11 | 11 | 13 | 7 | 16
  Fatigue | 18 | 19 | 22 | 24 | 23 | 23 | 16 | 26
  Fever (≥38°C) | 2 | 2 | 2 | 0 | 3 | 0 | 2 | 0
  Other | 15 | 11 | 7 | 10 | 13 | 12 | 10 | 12
  Stayed at home due to reaction | 3 | 2 | 3 | 2 | 6 | 3 | 4 | 5
  Analgesic antipyretic medication used | 14 | 11 | 7 | 9 | 11 | 10 | 8 | 10

ADVERSE EVENTS:
Time Frame: Through out the study period
Description: Post-injection solicited adverse events were collected from Day 1-7. Other AEs and SAEs were collected through out the study period (Day 1 to 6 months).
Groups:
- Adults (cTIV\cTIV) + (TIV\cTIV): Subjects(18-60 years of age) who previously received one dose of either cell-derived (cTIV) or egg derived (TIV) trivalent influenza vaccine received one dose of cTIV in this study, one year later.
- Adults (cTIV/TIV) + (TIV\TIV): Subjects (18-60 years of age) who previously received one dose of either cell-derived (cTIV) or egg derived (TIV) trivalent influenza vaccine received one dose of TIV in this study, one year later.
- Elderly (cTIV\cTIV) + (TIV\cTIV): Subjects(≥61 years of age) who previously received one dose of either cell-derived (cTIV) or egg derived (TIV) trivalent influenza vaccine received one dose of cTIV in this study, one year later.
Arm/Group | Adults (cTIV\cTIV) + (TIV\cTIV) | Adults (cTIV/TIV) + (TIV\TIV) | Elderly (cTIV\cTIV) + (TIV\cTIV) | Elderly (cTIV\TIV) + (TIV\TIV)
Serious Adverse Events (participants affected / at risk) | 9/533 | 4/534 | 23/571 | 30/597
Other Adverse Events (participants affected / at risk) | 188/533 | 172/534 | 140/571 | 148/597
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults (cTIV\cTIV) + (TIV\cTIV) (N=533) | Adults (cTIV/TIV) + (TIV\TIV) (N=534) | Elderly (cTIV\cTIV) + (TIV\cTIV) (N=571) | Elderly (cTIV\TIV) + (TIV\TIV) (N=597)
Acute myocardial infraction (Cardiac disorders) | 0 | 0 | 2 | 1
Adams stokes syndrome (Cardiac disorders) | 0 | 0 | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia paroxysmal (Cardiac disorders) | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Spilgelian hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Umblical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bronchitis acute (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis chronic (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Toe deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Blood electrolytes abnormal (Investigations) | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infraction (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Angineurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 0 | 1 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 0 | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0
Arteriosclerosis obliterans (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adults (cTIV\cTIV) + (TIV\cTIV) (N=533) | Adults (cTIV/TIV) + (TIV\TIV) (N=534) | Elderly (cTIV\cTIV) + (TIV\cTIV) (N=571) | Elderly (cTIV\TIV) + (TIV\TIV) (N=597)
Fatigue (General disorders) | 41 | 43 | 49 | 41
Injection site erythema (General disorders) | 59 | 66 | 46 | 35
Injection site induration (General disorders) | 35 | 31 | 24 | 17
Injection site haemorrhage (General disorders) | 26 | 24 | 23 | 33
Injection site pain (General disorders) | 115 | 91 | 48 | 40
Malaise (General disorders) | 48 | 43 | 49 | 39
Myalgia (Musculoskeletal and connective tissue disorders) | 40 | 42 | 36 | 20
Headache (Nervous system disorders) | 55 | 42 | 38 | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 16 | 31 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days